CLINICAL TRIAL: NCT01111123
Title: A Randomized, Double-blind Study to Evaluate the Efficacy of Ammonium Lactate Lotion 12% (Lac-hydrin®) and Halobetasol Propionate Ointment 0.05% (Ultravate®) in the Treatment and Maintenance of Psoriasis.
Brief Title: Ammonium Lactate Lotion 12% (Lac-hydrin®) and Halobetasol Propionate Ointment 0.05% (Ultravate®) in the Treatment and Maintenance of Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 08-1061 0001 01 DE
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; lac-hydrin; ammonium lactate; Ultravate; halobetasol propionate; weekend only application; topical therapy; topical corticosteroid; class I steroid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lac-Hydrin lotion twice daily everyday + Ultravate ointment twice daily on weekends only
  Interventions: Drug: Lac-Hydrin lotion (ammonium lactate lotion 12%) ; UItravate ointment (halobetasol propionate ointment 0.05%)
- 2 (Placebo Comparator): Lac-Hydrin lotion twice daily everyday + placebo ointment twice daily on weekends only
  Interventions: Drug: Lac-Hydrin lotion (ammonium lactate lotion 12%); placebo ointment

INTERVENTIONS:
Drug: Lac-Hydrin lotion (ammonium lactate lotion 12%) ; UItravate ointment (halobetasol propionate ointment 0.05%) — Steroid on weekends only group
  Arms: 1
Drug: Lac-Hydrin lotion (ammonium lactate lotion 12%); placebo ointment — Placebo on weekends only group
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the combinational use of ammonium lactate lotion 12% (Lac-Hydrin) and halobetasol propionate ointment 0.05% (Ultravate) is safe and effective in the initial treatment and long-term maintenance of psoriasis. Patients will use both medications continuously for two weeks and those who obtain a good improvement based on investigator clinical assessments will be randomized to Lac-Hydrin lotion twice daily every day with placebo ointment or Ultravate ointment twice daily on weekends only for up to 24 more weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, clinical trial assessing the efficacy of Ultravate ointment in combination with Lac-Hydrin lotion in the treatment of plaque psoriasis. In the first phase, patients will be treated for two weeks with combination therapy using Ultravate ointment twice daily along with Lac-Hydrin lotion twice daily. After two weeks, psoriasis plaques will be evaluated to test treatment efficacy. Those patients with a significant clinical improvement per investigator clinical assessments, will be randomized in a 1:1 fashion into a maintenance phase and receive Lac-Hydrin lotion twice daily everyday with placebo ointment or Ultravate ointment twice daily on weekends only. Continuous use of Ultravate ointment will be discontinued following two weeks of treatment in compliance with its FDA indication. Patients will be evaluated every 4 weeks (monthly) through the maintenance phase. The purpose of this second phase of the study is to investigate whether use of Ultravate on weekends only can minimize risk of plaque recurrence, maximize duration of therapeutic effect, while limiting the need for the use of long-term continuous topical corticosteroid treatment. As well, the second phase of the study is to investigate whether twice daily Lac-Hydrin lotion has an impact in maximizing the duration of therapeutic effect as well as minimizing local cutaneous side effects such as skin atrophy and telangiectasia. Part of this clinical study consists of the use of patient and self-assessment questionnaires and the use of non-identifying digital photography of target lesions. The hypothesis is that Ultravate ointment on weekends only will be statistically more efficacious at maintaining an excellent initial clinical response and its combination with Lac-Hydrin lotion will help to minimize any local cutaneous side effects as well as enhance its therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age and in good general health as confirmed by a medical history.
* Females of childbearing potential must have a negative urine pregnancy test on Day 1 and must agree to use adequate birth control methods during the entire study.
* A clear diagnosis of plaque psoriasis must have been previously established and the disease must have been present at least 6 months.
* Subjects must have lesions suitable for evaluating response to test agents. The severity of the disease at Day 1 must be rated at least 2 (Mild) for each of the key psoriasis characteristics (scaling, erythema, and plaque elevation).
* Subjects must be able to understand the requirements of the study, abide by the restrictions, and return for the required examinations. All subject must sign the statement of informed consent approved for the study.

Exclusion Criteria:

* Subjects who are pregnant (determined from a urine pregnancy test on Day 1).
* Subjects who are nursing.
* Subjects with known hypersensitivity to any components of the test medication.
* Subjects requiring any other medication (topical or systemic) that may affect the course of the disease during the study period (e.g. antibiotics, sedating antihistamines).
* Subjects using biologics or any other systemic treatment for psoriasis within 12 weeks of entering the study.
* Subjects using systemic corticosteroids within 28 days of entering the study; subjects using topical corticosteroids or other topical therapies (other than emollients) at any location on the body within 1 week of entering the study.
* Subjects with overt pre-existing telangiectasia or skin atrophy at intended treatment sites.
* Subjects who are using any medication or has any disease which in the judgment of the investigator will interfere with the conduct or interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Emer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Department of Dermatology, New York, New York, United States

REFERENCES:
- [Result] Emer JJ, Frankel A, Sohn A, Lebwohl M. A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Ammonium Lactate Lotion 12% and Halobetasol Propionate Ointment 0.05% in the Treatment and Maintenance of Psoriasis. J Clin Aesthet Dermatol. 2011 Feb;4(2):28-39. PMID 21386955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at the outpatient clinic of the MSSM Department of Dermatology Clinical Trials Center, in New York, New York, from January 2009 to March 2010. Recruitment was through: advertisements, referrals from the Dermatology Faculty Practice Associates, and through voluntary faculty and dermatology residents.
Pre-assignment Details: Patients who were pregnant/nursing, those on biological or other systemic treatments or other systemic treatments in previous three months, those on topical therapies other than emollients in the past one month, those with pre-existing overt atrophy/telangiectasia in treatment areas were excluded.
Groups:
- Lac-hydrin + Ultravate: Lac-Hydrin lotion twice daily everyday + Ultravate ointment twice daily on weekends only, for up to 24 weeks
- Lac Hydrin + Placebo: Lac-Hydrin lotion twice daily everyday + placebo ointment twice daily on weekends only, for up to 24 weeks
Period: Open- Label Phase
Arm/Group | Lac-hydrin + Ultravate | Lac Hydrin + Placebo
Started | 55 | 0
Completed | 41 | 0
Not Completed | 14 | 0
Not completed — Failed to be clear or almost cleared | 14 | 0
Period: Maintenance Phase
Arm/Group | Lac-hydrin + Ultravate | Lac Hydrin + Placebo
Started | 21 | 20
Completed | 21 | 18
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lac-hydrin + Ultravate | Lac Hydrin + Placebo | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Physical Global Assessment
Description: Physician global assessment (PGA) score - the physician's impression of the disease at a single time point rated as: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, and 5=very severe.
Time Frame: During the maintenance phase, from 2 weeks up to 26 weeks
Population: The primary endpoint was a change in PGA during the 24 weeks of the study in the intention-to-treat population (ITT).
Measure: Number; unit: participants
Groups:
- Ammonium Lactate + Ultravate: ammonium lactate twice daily everyday plus ultravte ointment twice daily on weekends only for up to 24 weeks
- Ammoium Lactate + Placebo: ammonium lactate twice daily everyday plus placebo ointment twice daily weekends only
Arm/Group | Ammonium Lactate + Ultravate | Ammoium Lactate + Placebo
Number analyzed (Participants) | 21 | 20
participants
  Category 0 or 1 | 12 | 0
  Category ≥ 2 | 9 | 20
Statistical Analysis 1: Comparison: Ammonium Lactate + Ultravate vs Ammoium Lactate + Placebo; Probabilities of PGA not worsening were estimated using the Kaplan-Meier product limit method with a comparison between treatment group survival curves evaluated by the log-rank test statistic. The Cox proportional hazards model was used to estimate the hazard ratio for worsening of PGA (equivalent to a relative risk adjusted for follow-up time) and a corresponding 95-percent confidence interval; Test type: Superiority or Other; p < 0.05, Log Rank — CI of 95%

2. Secondary Outcome: Signs of Psoriasis, Atrophy or Telangiectasis
Description: Signs of psoriasis (erythema, induration, and scale) - physician's assessment of the severity of each of the three key characteristics of psoriatic lesions rated as: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, and 5=very severe, combined into one score.
Time Frame: During the maintenance phase, from 2 weeks up to 26 weeks
Population: The primary endpoint was a change in PGA during the 24 weeks of the study in the ITT.
Measure: Number; unit: participants
Groups:
- Lac-hydrin + Ultravate: ammonium lactate twice daily everyday + ultravate twice daily weekends only
- Lac-hydrin + Placebo: lac hydrin twice daily everyday plus placebo ointment twice daily weekends only
Arm/Group | Lac-hydrin + Ultravate | Lac-hydrin + Placebo
Number analyzed (Participants) | 21 | 20
participants
  category 0 or 1 | 12 | 0
  category ≥ 2 | 9 | 20
Statistical Analysis 1: Comparison: Lac-hydrin + Ultravate vs Lac-hydrin + Placebo; Secondary outcomes, including subject self-assessment and signs of psoriasis ratings, were analyzed as continuous dependent variables in these statistical models. Mixed modeling analysis of covariance (ANCOVA) was used to compare the relationships between psoriasis symptoms over time in the placebo and steroid treatment groups; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded up to the study total of 26 weeks. No follow-up visits were conducted after study treatment concluded.
Description: There were no reported AEs, including serious AEs, related to study medication throughout the study.
Arm/Group | Lac-hydrin + Ultravate | Lac Hydrin + Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
The maintenance phase did not have a long enough study duration to capture clinically significant changes in disease status in the steroid group since >50 percent of the patients at the end of the 24 weeks still remained in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No